CLINICAL TRIAL: NCT04707963
Title: Peanut Protein Supplementation to Augment Muscle Growth and Improve Markers of Muscle Quality and Health in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: Edward Via College of Osteopathic Medicine-Auburn (Unknown); The Peanut Institute (Other)
Responsible Party: Principal Investigator, Andrew Fruge, Assistant Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 19-249B
Record Dates: First submitted 2021-01-10; First posted 2021-01-13 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Sarcopenia
Keywords: resistance training; muscle hypertrophy; muscle quality
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Intervention group will receive the supplement during the study period and the wait-listed control group will receive the supplement after the study period. Both groups will participate in resistance training during the 10 week period
Who Masked: Investigator, Outcomes Assessor
Masking Description: PI and Co-Is will be blind to participant randomization. One study staff member will be responsible for administering the supplements to participants per randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): Participants will complete 10 weeks of twice-weekly whole body resistance training. Peanut protein powder (72g/day) will be provided for daily consumption during the study period
  Interventions: Dietary Supplement: Peanut protein powder; Behavioral: Full body resistance training
- Wait-list Control Group (Active Comparator): Participants will complete 10 weeks of twice-weekly whole body resistance training. Peanut protein powder will be provided after the study period
  Interventions: Behavioral: Full body resistance training

INTERVENTIONS:
Dietary Supplement: Peanut protein powder — Peanut protein powder will be provided to participants who will be instructed to consume 72g daily, mixed with water
  Arms: Immediate Intervention Group
Behavioral: Full body resistance training — Participants will undergo supervised resistance training two times per week (5 exercises, 3 sets of 8-12 repetitions per set)

SUMMARY:
This study will evaluate the adaptations in skeletal muscle that occur in response to 10 weeks of weight training with or without peanut protein supplementation in untrained men and women ages 18-30

DETAILED DESCRIPTION:
This is a two-phase study using both novel and conventional methods to assess how PP supplementation affects muscle tissue in young adults who engage in resistance training. These two phases will be conducted as part of a 10-week randomized controlled trial in which men and women aged 18-30 years (n=40), will be stratified by gender and randomized to a resistance training intervention (whole body, two days per week) with PP powder (72g daily; n=10 males, n=10 females) provided during the intervention (immediate group, IG) or after the intervention (wait-list control, WLC, n=10 males, n=10 females). The aims of this study are to determine the acute (deuterium oxide tracer) and chronic (peripheral quantitative computed tomography) effects of PP during resistance training on skeletal muscle myofibrillar protein synthesis rates, changes in skeletal muscle size and quality, changes in whole and appendicular body composition (dual energy x-ray absorptiometry), changes in inflammatory markers and the fecal microbiome.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (body mass/height squared) less than 35 kg/m2
* resting blood pressure averaging less than 140/90 mmHg (with or without medication)

Exclusion Criteria:

* known peanut allergy
* actively participating in resistance training for more than 2 days/week
* any known overt cardiovascular or metabolic disease
* metal implants that will interfere with x-ray procedures
* medically necessary radiation exposure in the last six months (except dental x-ray)
* any medical condition that would contradict participating in an exercise program, giving blood or donating a skeletal muscle biopsy (i.e. blood clotting disorder or taking blood thinners)
* pregnant or trying to become pregnant

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-02-06 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change in acute myofibrillar protein synthesis rates | 24 hours
  Change in right leg vastus lateralis myofibrillar protein synthesis rates using the integrated deuterium oxide technique from biopsies immediately before and 24 hours after resistance exercise
  Change in right leg vastus lateralis myofibrillar protein synthesis rates using the integrated deuterium oxide technique from biopsies immediately before and 24 hours after resistance exercise
Change in mid-thigh skeletal muscle area and quality | 0-10 weeks
  Peripheral quantitative computed tomography (pQCT) cross-sectional image of mid-right thigh assessed for overall muscle density (mg/cm^3)

SECONDARY OUTCOMES:
Change in appendicular lean mass | 0-10 weeks
  Change in lean mass (kg) of limbs as measured by dual energy x-ray absorptiometry (DXA)
Change in Type I and II Muscle Fiber Cross-Sectional Area | 0-10 weeks
  Muscle biopsy immunofluorescent staining for determination of type I and type II muscle fiber cross sectional area (fCSA) as a cellular determinant of skeletal muscle hypertrophy
Change in leg extensor isokinetic dynamometry | 0-10 weeks
  maximal isokinetic right leg extensions on an isokinetic dynamometer (BioDex)
Change in fecal microbiome composition | 0-10 weeks
  alpha- and beta-diversity of 16S bacterial rDNA

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Roberts, PhD, Principal Investigator — Associate Professor
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified anthropometric, physiological, biological and performance data may be requested

REFERENCES:
- [Derived] Sexton CL, Smith MA, Smith KS, Osburn SC, Godwin JS, Ruple BA, Hendricks AM, Mobley CB, Goodlett MD, Fruge AD, Young KC, Roberts MD. Effects of Peanut Protein Supplementation on Resistance Training Adaptations in Younger Adults. Nutrients. 2021 Nov 9;13(11):3981. doi: 10.3390/nu13113981. PMID 34836236